CLINICAL TRIAL: NCT01475734
Title: A Single-site, Randomized, Double-blind, Placebo-controlled, Parallel-group, Stepped Glucose Clamp Study to Assess the Effects of Albiglutide on Counter-regulatory Hormone Responses and Recovery From Hypoglycemia in Subjects With Type 2 Diabetes Mellitus.
Brief Title: Albiglutide Glucose Clamp Study in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 108372
Record Dates: First submitted 2011-11-17; First posted 2011-11-21 (Estimated); Results first posted 2014-05-16 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: glucose clamp; hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypoglycemia | interventions — rGLP-1 protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- albiglutide (Active Comparator): single dose of albiglutide
  Interventions: Biological: albiglutide
- placebo (Placebo Comparator): single dose of placebo
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: albiglutide — subcutaneous injection
  Arms: albiglutide
Biological: placebo — subcutaneous injection
  Arms: placebo

SUMMARY:
This is a stepped glucose clamp study designed to investigate the effect of treatment with albiglutide on counter-regulatory hormone responses and recovery from hypoglycemia in subjects with Type 2 diabetes mellitus. A single dose of albiglutide or placebo will be given prior to a stepped hyper- and hypoglycemic clamp. The goal of this study is to demonstrate that albiglutide increases insulin secretion and decreases glucagon levels in a glucose-dependent manner.

DETAILED DESCRIPTION:
This is a Phase II, single-site, randomized, double-blind, parallel-group, placebo-controlled, stepped glucose clamp study designed to investigate the effect of treatment with albiglutide on counter-regulatory hormone responses and recovery from hypoglycemia in subjects with Type 2 diabetes mellitus. A single dose of albiglutide or placebo will be given 3 days before employing a stepped hyper- and hypoglycemic clamp. The goal of this study is to demonstrate that albiglutide increases insulin secretion and decreases glucagon levels in a glucose-dependent manner. In particular, this study is being conducted to ensure that albiglutide does not impair counter-regulatory responses during hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

* Historical diagnosis of type 2 diabetes mellitus for at least 6 months and less than 10 years before Screening
* HbA1c <10% at Screening for subjects who do not require washout of existing OAD or <9% at Screening for subjects who do require washout from existing OAD
* Body mass index in range 28 kg/m2 to40 kg/m2

Exclusion Criteria:

* History of pancreatitis or current ongoing symptomatic biliary disease or pancreatitis
* History of significant gastrointestinal surgery,
* History of significant cardiovascular disease
* History of a seizure disorder
* Documented hypertension or hypotension
* Use of oral antidiabetic agents, except for metformin, within 14 days before investigational product administration.
* Current hepatic disease or abnormal liver function tests
* Positive test result for hepatitis B, hepatitis C, or human immunodeficiency virus infection 1 or 2
* History of regular alcohol consumption (exceeding 7 drinks/week for women or 14 drinks/week for men)
* Female subject is pregnant (confirmed by laboratory testing), lactating, or less than 6 weeks postpartum
* Known allergy to any GLP-1 analog or excipients of albiglutide, Baker's yeast, or insulin
* History of type 1 diabetes,
* Prior exposure to GLP-1 agents, including albiglutide
* Blood donation over 500 mL within 8 weeks before Screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2011-12; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Chula Vista, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Young MA, Wald JA, Matthews JE, Scott R, Hodge RJ, Zhi H, Reinhardt RR. Clinical pharmacology of albiglutide, a GLP-1 receptor agonist. Postgrad Med. 2014 Nov;126(7):84-97. doi: 10.3810/pgm.2014.11.2836. PMID 25387217
- [Derived] Hompesch M, Jones-Leone A, Carr MC, Matthews J, Zhi H, Young M, Morrow L, Reinhardt RR. Albiglutide does not impair the counter-regulatory hormone response to hypoglycaemia: a randomized, double-blind, placebo-controlled, stepped glucose clamp study in subjects with type 2 diabetes mellitus. Diabetes Obes Metab. 2015 Jan;17(1):82-90. doi: 10.1111/dom.12398. Epub 2014 Oct 26. PMID 25263215
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 108372 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 108372 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 108372 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 108372 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 108372 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 108372 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 108372 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible participants entered a 1-week Screening Period, a 2-week Run-in/Stabilization Period, a 4-day Treatment Period for the evaluation of efficacy and safety, and an 8-week post-treatment Follow-up Period. A total of 45 participants were screened, 44 were randomized, and 41 completed the study.
Groups:
- Albiglutide 50 mg: Participants received a single dose of albiglutide (50 milligrams [mg]) subcutaneously 3 days before employing a stepped hyper- and hypoglycemic clamp with glucose plateaus of 9.0, 5.0, 4.0, 3.3, and 2.8 millimoles per liter (mmol/L) (162, 90, 72, 59, and 50.4 milligrams per deciliter [mg/dL], respectively). Glucose and insulin infusions were included as part of the clamp procedure.
- Placebo: Participants received a single dose of matching placebo (50 mg) subcutaneously 3 days before employing a stepped hyper- and hypoglycemic clamp with glucose plateaus of 9.0, 5.0, 4.0, 3.3, and 2.8 mmol/L (162, 90, 72, 59, and 50.4 mg/dL, respectively). Glucose and insulin infusions were included as part of the clamp procedure.
Period: Overall Study
Arm/Group | Albiglutide 50 mg | Placebo
Started | 22 | 22
Completed | 20 | 21
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Albiglutide 50 mg | Placebo | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.9 (6.86) | 48.4 (9.32) | 49.1 (8.12)
Gender [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 10 | 10 | 20
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 1 | 5 | 6
  White - Arabic/North African Heritage | 0 | 1 | 1
  White - White/Caucasian/European Heritage | 20 | 14 | 34
  Hispanic | 0 | 1 | 1
  Mexican | 1 | 0 | 1
  Persian | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Glucagon Concentration (Nanomoles Per Liter [Nmol/L]) During the Hypoglycemic Periods of the Glucose Clamp Procedure
Description: Plasma glucagon levels were measured for the estimation of glucagon secretion during the hypoglycemic periods. Glucagon response was measured at each clamped glucose concentration: 9 millimoles per liter (mmol/L) (0 hour [hr], 1hr, 1 hr 15 minutes [min]), 5 mmol/L (1 hr 45 min, 2 hr), 4 mmol/L (2 hr 45 min, 3 hr), 3.3 mmol/L (3 hr 30 min, 3 hr 45 min), and 2.8 mmol/L (4 hr 15 min, 4 hr 30 min), and clamp released (4 hr 45 min, 5 hr, 5 hr 15 min, 5 hr 30 min). Repeated-measures analysis of variance was performed on non-transformed pharmacodynamic parameters using a model with treatment, time, and treatment-by-time as fixed effects, and participant as a random effect. Values below the lower limit of quantification (0.03780 nmol/L) were set to the quantification limit for summary.
Time Frame: Day 4
Population: Pharmacodynamic (PD) Population: all participants who received 1 dose of albiglutide or placebo, had a Baseline assessment, and had at least 1 post-Baseline assessment of the primary endpoint (glucagon) during the clamp procedure. PD Population participants were analyzed according to randomly assigned treatment.
Measure: Geometric Mean (Standard Deviation); unit: Nanomoles per liter (nmol/L)
Arm/Group | Albiglutide 50 mg | Placebo
Number analyzed (Participants) | 20 | 21
Nanomoles per liter (nmol/L)
  0 hr, n=20, 21 | 0.03780 (1.000000) | 0.03805 (1.030606)
  1 hr, n=20, 21 | 0.03780 (1.000000) | 0.03780 (1.000000)
  1 hr 15 min, n=20, 21 | 0.03783 (1.003528) | 0.03780 (1.000000)
  1 hr 45 min, n=20, 21 | 0.03780 (1.000000) | 0.03780 (1.000000)
  2 hr, n=20, 20 | 0.03805 (1.029775) | 0.03780 (1.000000)
  2 hr 45 min, n=20, 21 | 0.03876 (1.090802) | 0.03780 (1.000000)
  3 hr, n=20, 21 | 0.03808 (1.024552) | 0.03780 (1.000000)
  3 hr 30 min, n=20, 21 | 0.04296 (1.203416) | 0.03922 (1.127202)
  3 hr 45 min, n=20, 21 | 0.04072 (1.146327) | 0.03893 (1.086818)
  4 hr 15 min, n=20, 21 | 0.03976 (1.152056) | 0.04094 (1.192380)
  4 hr 30 min, n=20, 21 | 0.03899 (1.105904) | 0.04000 (1.146223)
  4 hr 45 min, n=20, 21 | 0.03936 (1.102107) | 0.03958 (1.116342)
  5 hr, n=20, 21 | 0.03780 (1.000000) | 0.03814 (1.042285)
  5 hr 15 min, n=20, 21 | 0.03809 (1.034545) | 0.03780 (1.000000)
  5 hr 30 min, n=20, 21 | 0.03780 (1.000000) | 0.03780 (1.000000)
Statistical Analysis 1: Comparison: Albiglutide 50 mg vs Placebo; Test type: Superiority or Other; p = 0.791, ANOVA; Ratio = 0.993, 95% CI 2-sided [0.946 to 1.043] — The estimated value represents the ratio of geometric least squares means (albiglutide 50 mg) to placebo at 0 hr
Statistical Analysis 2: Comparison: Albiglutide 50 mg vs Placebo; Test type: Superiority or Other; p > 0.999, ANOVA; Ratio = 1.000, 95% CI 2-sided [0.952 to 1.050] — The estimated value represents the ratio of geometric least squares means (albiglutide 50 mg) to placebo at 1 hr
Statistical Analysis 3: Comparison: Albiglutide 50 mg vs Placebo; Test type: Superiority or Other; p = 0.975, ANOVA; Ratio = 1.001, 95% CI 2-sided [0.953 to 1.051] — The estimated value represents the ratio of geometric least squares means (albiglutide 50 mg) to placebo at 1 hr 15 min
Statistical Analysis 4: Comparison: Albiglutide 50 mg vs Placebo; Test type: Superiority or Other; p > 0.999, ANOVA; Ratio = 1.000, 95% CI 2-sided [0.952 to 1.050] — The estimated value represents the ratio of geometric least squares means (albiglutide 50 mg) to placebo at 1 hr 45 min
Statistical Analysis 5: Comparison: Albiglutide 50 mg vs Placebo; Test type: Superiority or Other; p = 0.908, ANOVA; Ratio = 1.003, 95% CI 2-sided [0.955 to 1.053] — The estimated value represents the ratio of geometric least squares means (albiglutide 50 mg) to placebo at 2 hr
Statistical Analysis 6: Comparison: Albiglutide 50 mg vs Placebo; Test type: Superiority or Other; p = 0.312, ANOVA; Ratio = 1.025, 95% CI 2-sided [0.977 to 1.077] — The estimated value represents the ratio of geometric least squares means (albiglutide 50 mg) to placebo at 2 hr 45 min
Statistical Analysis 7: Comparison: Albiglutide 50 mg vs Placebo; Test type: Superiority or Other; p = 0.763, ANOVA; Ratio = 1.008, 95% CI 2-sided [0.960 to 1.058] — The estimated value represents the ratio of geometric least squares means (albiglutide 50 mg) to placebo at 3 hr
Statistical Analysis 8: Comparison: Albiglutide 50 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANOVA; Ratio = 1.095, 95% CI 2-sided [1.043 to 1.150] — The estimated value represents the ratio of geometric least squares means (albiglutide 50 mg) to placebo at 3 hr 30 min
Statistical Analysis 9: Comparison: Albiglutide 50 mg vs Placebo; Test type: Superiority or Other; p = 0.070, ANOVA; Ratio = 1.046, 95% CI 2-sided [0.996 to 1.098] — The estimated value represents the ratio of geometric least squares means (albiglutide 50 mg) to placebo at 3 hr 45 min
Statistical Analysis 10: Comparison: Albiglutide 50 mg vs Placebo; Test type: Superiority or Other; p = 0.238, ANOVA; Ratio = 0.971, 95% CI 2-sided [0.925 to 1.020] — The estimated value represents the ratio of geometric least squares means (albiglutide 50 mg) to placebo at 4 hr 15 min
Statistical Analysis 11: Comparison: Albiglutide 50 mg vs Placebo; Test type: Superiority or Other; p = 0.298, ANOVA; Ratio = 0.975, 95% CI 2-sided [0.928 to 1.023] — The estimated value represents the ratio of geometric least squares means (albiglutide 50 mg) to placebo at 4 hr 30 min
Statistical Analysis 12: Comparison: Albiglutide 50 mg vs Placebo; Test type: Superiority or Other; p = 0.821, ANOVA; Ratio = 0.994, 95% CI 2-sided [0.947 to 1.044] — The estimated value represents the ratio of geometric least squares means (albiglutide 50 mg) to placebo at 4 hr 45 min
Statistical Analysis 13: Comparison: Albiglutide 50 mg vs Placebo; Test type: Superiority or Other; p = 0.715, ANOVA; Ratio = 0.991, 95% CI 2-sided [0.944 to 1.040] — The estimated value represents the ratio of geometric least squares means (albiglutide 50 mg) to placebo at 5 hr
Statistical Analysis 14: Comparison: Albiglutide 50 mg vs Placebo; Test type: Superiority or Other; p = 0.759, ANOVA; Ratio = 1.008, 95% CI 2-sided [0.960 to 1.058] — The estimated value represents the ratio of geometric least squares means (albiglutide 50 mg) to placebo at 5 hr 15 min
Statistical Analysis 15: Comparison: Albiglutide 50 mg vs Placebo; Test type: Superiority or Other; p > 0.999, ANOVA; Ratio = 1.000, 95% CI 2-sided [0.952 to 1.050] — The estimated value represents the ratio of geometric least squares means (albiglutide 50 mg) to placebo at 5 hr 30 min

2. Secondary Outcome: Insulin Secretion Rate (Measured by Mathematical Analysis of C-peptide Concentrations) During the Glucose Clamp Period
Description: The insulin secretion rate (ISR) was estimated by the deconvolution of peripheral C-peptide concentrations using a 2-compartment model that utilizes population C-peptide kinetic parameters. ISR was measured at 1 hr, 1 hr 15 min, 1 hr 45 min, 2 hr, 2 hr 45 min, 3 hr, 3 hr 30 min, 3 hr 45 min, 4 hr 15 min, and 4 hr 30 min. Repeated-measures analysis of variance was performed on insulin secretion rate using a model with treatment, time, and treatment-by-time as fixed effects, and participant as a random effect.
Time Frame: Day 4
Population: Pharmacodynamic Population
Measure: Mean (Standard Deviation); unit: Milliunits per hour (mU/hr)
Arm/Group | Albiglutide 50 mg | Placebo
Number analyzed (Participants) | 20 | 21
Milliunits per hour (mU/hr)
  1 hr | 0.22992 (0.175853) | 0.15487 (0.111490)
  1 hr 15 min | 0.32088 (0.262743) | 0.22083 (0.143504)
  1 hr 45 min | 0.02309 (0.155010) | -0.00873 (0.052095)
  2 hr | 0.14532 (0.152512) | 0.08063 (0.105769)
  2 hr 45 min | 0.01411 (0.038786) | 0.02484 (0.030589)
  3 hr | 0.03145 (0.042047) | 0.04148 (0.038344)
  3 hr 30 min | -0.02053 (0.047566) | -0.00507 (0.033461)
  3 hr 45 min | 0.01197 (0.015914) | 0.01878 (0.014128)
  4 hr 15 min | 0.00892 (0.017889) | 0.01401 (0.009209)
  4 hr 30 min | 0.01868 (0.011193) | 0.02254 (0.003796)

3. Secondary Outcome: Epinephrine Values During the Glucose Clamp Period
Description: Epinephrine levels were measured at all stages of glycemia during the glucose clamp period. Epinephrine levels were measured at each clamped glucose concentration: 9 millimoles per liter (mmol/L) (0 hour [hr], 1hr, 1 hr 15 minutes [min]), 5 mmol/L (1 hr 45 min, 2 hr), 4 mmol/L (2 hr 45 min, 3 hr), 3.3 mmol/L (3 hr 30 min, 3 hr 45 min), and 2.8 mmol/L (4 hr 15 min, 4 hr 30 min), and clamp released (4 hr 45 min, 5 hr, 5 hr 15 min, 5 hr 30 min). Repeated-measures analysis of variance was performed on log-transformed pharmacodynamic parameters using a model with treatment, time, and treatment-by-time as fixed effects, and participant as a random effect. Values below the lower limit of quantification were set to the quantification limit for summary.
Time Frame: Day 4
Population: Pharmacodynamic Population. Different participants may have been analyzed at different time points (reflected by n=X, X in the category titles), so the overall number of participants analyzed reflects everyone in the Pharmacodynamic Population.
Measure: Geometric Mean (Standard Deviation); unit: Nanograms per liter (ng/L)
Arm/Group | Albiglutide 50 mg | Placebo
Number analyzed (Participants) | 20 | 21
Nanograms per liter (ng/L)
  0 hr, n=19, 20 | 56.9 (1.38) | 59.4 (1.49)
  1 hr, n=19, 18 | 60.7 (1.78) | 61.2 (1.52)
  1 hr 15 min, n=18, 19 | 57.8 (1.37) | 59.9 (1.48)
  1 hr 45 min, n=20, 21 | 69.1 (1.38) | 70.1 (1.52)
  2 hr, n=20, 20 | 73.2 (1.44) | 81.5 (1.61)
  2 hr 45 min, n=20, 21 | 183.9 (1.89) | 159.2 (1.82)
  3 hr, n=19, 21 | 187.1 (1.81) | 171.1 (1.97)
  3 hr 30 min, n=19, 21 | 429.2 (1.73) | 372.3 (1.97)
  3 hr 45 min, n=20, 21 | 410.3 (1.93) | 318.8 (2.21)
  4 hr 15 min, n=20, 21 | 568.3 (1.93) | 519.5 (1.92)
  4 hr 30 min, n=20, 21 | 608.7 (1.80) | 505.6 (2.18)
  4 hr 45 min, n=20, 21 | 477.1 (1.97) | 395.4 (2.15)
  5 hr, n=20, 21 | 246.6 (2.04) | 225.9 (2.01)
  5 hr 15 min, n=20, 21 | 172.4 (2.14) | 154.4 (1.67)
  5 hr 30 min, n=20, 21 | 132.5 (1.85) | 118.2 (1.62)

4. Secondary Outcome: Norepinephrine Values During the Glucose Clamp Period
Description: Norepinephrine levels were measured at all stages of glycemia during the glucose clamp period. Epinephrine levels were measured at each clamped glucose concentration: 9 millimoles per liter (mmol/L) (0 hour [hr], 1hr, 1 hr 15 minutes [min]), 5 mmol/L (1 hr 45 min, 2 hr), 4 mmol/L (2 hr 45 min, 3 hr), 3.3 mmol/L (3 hr 30 min, 3 hr 45 min), and 2.8 mmol/L (4 hr 15 min, 4 hr 30 min), and clamp released (4 hr 45 min, 5 hr, 5 hr 15 min, 5 hr 30 min). Repeated-measures analysis of variance was performed on log-transformed pharmacodynamic parameters using a model with treatment, time, and treatment-by-time as fixed effects, and participant as a random effect. Values below the lower limit of quantification were set to the quantification limit for summary.
Time Frame: Day 4
Population: as for outcome 3
Measure: Geometric Mean (Standard Deviation); unit: Nanograms per liter (ng/L)
Arm/Group | Albiglutide 50 mg | Placebo
Number analyzed (Participants) | 20 | 21
Nanograms per liter (ng/L)
  0 hr, n=20, 21 | 340.6 (1.45) | 357.0 (1.44)
  1 hr, n=20, 21 | 347.1 (1.44) | 360.9 (1.55)
  1 hr 15 min, n=19, 21 | 382.3 (1.40) | 376.2 (1.57)
  1 hr 45 min, n=20, 21 | 347.7 (1.48) | 424.6 (1.48)
  2 hr, n=20, 20 | 346.3 (1.42) | 382.5 (1.33)
  2 hr 45 min, n=20, 21 | 425.5 (1.51) | 421.2 (1.53)
  3 hr, n=20, 21 | 425.0 (1.58) | 411.9 (1.50)
  3 hr 30 min, n=20, 21 | 543.2 (1.59) | 519.2 (1.55)
  3 hr 45 min, n=20, 21 | 537.5 (1.57) | 447.5 (1.53)
  4 hr 15 min, n=20, 21 | 624.0 (1.55) | 618.0 (1.40)
  4 hr 30 min, n=20, 21 | 649.5 (1.57) | 622.2 (1.44)
  4 hr 45 min, n=20, 21 | 605.0 (1.63) | 605.8 (1.38)
  5 hr , n=20, 21 | 508.4 (1.61) | 485.4 (1.30)
  5 hr 15 min, n=20, 21 | 511.3 (1.56) | 464.4 (1.42)
  5 hr 30 min, n=20, 21 | 469.4 (1.50) | 444.7 (1.42)

5. Secondary Outcome: Growth Hormone Values During the Glucose Clamp Period
Description: Growth hormone levels were measured at all stages of glycemia during the glucose clamp period. Epinephrine levels were measured at each clamped glucose concentration: 9 millimoles per liter (mmol/L) (0 hour [hr], 1hr, 1 hr 15 minutes [min]), 5 mmol/L (1 hr 45 min, 2 hr), 4 mmol/L (2 hr 45 min, 3 hr), 3.3 mmol/L (3 hr 30 min, 3 hr 45 min), and 2.8 mmol/L (4 hr 15 min, 4 hr 30 min), and clamp released (4 hr 45 min, 5 hr, 5 hr 15 min, 5 hr 30 min). Repeated-measures analysis of variance was performed on log-transformed pharmacodynamic parameters using a model with treatment, time, and treatment-by-time as fixed effects, and participant as a random effect. Values below the lower limit of quantification were set to the quantification limit for summary.
Time Frame: Day 4
Population: as for outcome 3
Measure: Geometric Mean (Standard Deviation); unit: Micrograms per liter (µg/L)
Arm/Group | Albiglutide 50 mg | Placebo
Number analyzed (Participants) | 20 | 21
Micrograms per liter (µg/L)
  0 hr, n=20, 21 | 0.29 (3.093) | 0.26 (2.875)
  1 hr, n=20, 21 | 0.17 (2.170) | 0.23 (2.791)
  1 hr 15 min, n=20, 21 | 0.16 (2.294) | 0.26 (2.722)
  1 hr 45 min, n=20, 21 | 0.34 (3.160) | 0.41 (3.729)
  2 hr, n=20, 20 | 0.60 (3.343) | 0.59 (4.696)
  2 hr 45 min, n=20, 21 | 2.44 (2.910) | 2.25 (3.080)
  3 hr, n=20, 21 | 3.16 (2.641) | 3.50 (1.971)
  3 hr 30 min, n=20, 21 | 4.83 (1.764) | 4.81 (1.832)
  3 hr 45 min, n=20, 21 | 4.36 (1.868) | 4.61 (1.819)
  4 hr 15 min, n=20, 21 | 3.59 (1.864) | 4.34 (1.515)
  4 hr 30 min, n=20, 21 | 3.39 (1.722) | 4.16 (1.496)
  4 hr 45 min, n=20, 21 | 3.41 (1.703) | 3.93 (1.606)
  5 hr, n=20, 21 | 2.55 (1.778) | 2.99 (1.812)
  5 hr 15 min, n=20, 21 | 1.77 (2.030) | 1.93 (1.945)
  5 hr 30 min, n=20, 21 | 1.07 (1.906) | 1.14 (2.024)

6. Secondary Outcome: Insulin Values During the Glucose Clamp Period
Description: Insulin levels were measured at all stages of glycemia during the glucose clamp period. Epinephrine levels were measured at each clamped glucose concentration: 9 millimoles per liter (mmol/L) (0 hour [hr], 1hr, 1 hr 15 minutes [min]), 5 mmol/L (1 hr 45 min, 2 hr), 4 mmol/L (2 hr 45 min, 3 hr), 3.3 mmol/L (3 hr 30 min, 3 hr 45 min), and 2.8 mmol/L (4 hr 15 min, 4 hr 30 min), and clamp released (4 hr 45 min, 5 hr, 5 hr 15 min, 5 hr 30 min). Repeated-measures analysis of variance was performed on log-transformed pharmacodynamic parameters using a model with treatment, time, and treatment-by-time as fixed effects, and participant as a random effect. Values below the lower limit of quantification were set to the quantification limit for summary.
Time Frame: Day 4
Population: as for outcome 3
Measure: Geometric Mean (Standard Deviation); unit: Picomoles per liter (pmol/L)
Arm/Group | Albiglutide 50 mg | Placebo
Number analyzed (Participants) | 20 | 21
Picomoles per liter (pmol/L)
  0 hr, n=20, 21 | 140.5 (1.60) | 102.4 (1.50)
  1 hr, n=20, 21 | 297.5 (2.11) | 183.6 (2.07)
  1 hr 15 min, n=20, 21 | 385.9 (2.14) | 270.9 (1.84)
  1 hr 45 min, n=20, 21 | 250.6 (2.03) | 207.4 (2.20)
  2 hr, n=20, 20 | 437.4 (2.01) | 357.3 (1.81)
  2 hr 45 min, n=20, 21 | 298.3 (2.05) | 191.9 (2.52)
  3 hr, n=20, 21 | 680.2 (2.10) | 438.7 (2.25)
  3 hr 30 min, n=20, 21 | 677.1 (2.34) | 488.0 (2.33)
  3 hr 45 min, n=20, 21 | 1000.6 (2.66) | 861.2 (2.01)
  4 hr 15 min, n=20, 21 | 1738.7 (2.09) | 887.9 (2.91)
  4 hr 30 min, n=20, 21 | 1057.8 (3.60) | 758.1 (2.27)
  4 hr 45 min, n=20, 21 | 203.0 (2.62) | 115.5 (2.55)
  5 hr, n=20, 21 | 121.7 (2.39) | 75.6 (2.37)
  5 hr 15 min, n=20, 21 | 99.5 (2.05) | 69.6 (2.35)
  5 hr 30 min, n=20, 21 | 94.0 (2.02) | 65.1 (2.15)

7. Secondary Outcome: Cortisol Values During the Glucose Clamp Period
Description: Cortisol levels were measured at all stages of glycemia during the glucose clamp period. Epinephrine levels were measured at each clamped glucose concentration: 9 millimoles per liter (mmol/L) (0 hour [hr], 1hr, 1 hr 15 minutes [min]), 5 mmol/L (1 hr 45 min, 2 hr), 4 mmol/L (2 hr 45 min, 3 hr), 3.3 mmol/L (3 hr 30 min, 3 hr 45 min), and 2.8 mmol/L (4 hr 15 min, 4 hr 30 min), and clamp released (4 hr 45 min, 5 hr, 5 hr 15 min, 5 hr 30 min). Repeated-measures analysis of variance was performed on log-transformed pharmacodynamic parameters using a model with treatment, time, and treatment-by-time as fixed effects, and participant as a random effect. Values below the lower limit of quantification were set to the quantification limit for summary.
Time Frame: Day 4
Population: as for outcome 3
Measure: Geometric Mean (Standard Deviation); unit: Nanomoles per liter (nmol/L)
Arm/Group | Albiglutide 50 mg | Placebo
Number analyzed (Participants) | 20 | 21
Nanomoles per liter (nmol/L)
  0 hr, n=20, 21 | 260.9 (2.05) | 282.9 (1.46)
  1 hr, n=20, 21 | 208.9 (2.05) | 250.5 (1.23)
  1 hr 15 min, n=20, 21 | 207.4 (2.04) | 272.3 (1.27)
  1 hr 45 min, n=20, 21 | 233.2 (2.04) | 230.2 (1.37)
  2 hr, n=20, 20 | 231.0 (2.04) | 230.7 (1.38)
  2 hr 45 min, n=20, 21 | 273.9 (1.88) | 290.4 (1.59)
  3 hr, n=20, 21 | 392.1 (1.50) | 344.0 (1.51)
  3 hr 30 min, n=20, 21 | 597.0 (1.28) | 534.7 (1.36)
  3 hr 45 min, n=20, 21 | 667.7 (1.20) | 583.0 (1.26)
  4 hr 15 min, n=20, 21 | 746.4 (1.21) | 674.0 (1.19)
  4 hr 30 min, n=20, 21 | 758.2 (1.20) | 705.2 (1.18)
  4 hr 45 min, n=20, 21 | 780.0 (1.18) | 712.0 (1.21)
  5 hr, n=20, 21 | 718.9 (1.32) | 673.3 (1.24)
  5 hr 15 min, n=20, 21 | 703.4 (1.20) | 626.8 (1.28)
  5 hr 30 min, n=20, 21 | 646.4 (1.25) | 569.0 (1.29)

8. Secondary Outcome: C-peptide Values During the Glucose Clamp Period
Description: C-peptide levels were measured at all stages of glycemia during the glucose clamp period. Epinephrine levels were measured at each clamped glucose concentration: 9 millimoles per liter (mmol/L) (0 hour [hr], 1hr, 1 hr 15 minutes [min]), 5 mmol/L (1 hr 45 min, 2 hr), 4 mmol/L (2 hr 45 min, 3 hr), 3.3 mmol/L (3 hr 30 min, 3 hr 45 min), and 2.8 mmol/L (4 hr 15 min, 4 hr 30 min), and clamp released (4 hr 45 min, 5 hr, 5 hr 15 min, 5 hr 30 min). Repeated-measures analysis of variance was performed on log-transformed pharmacodynamic parameters using a model with treatment, time, and treatment-by-time as fixed effects, and participant as a random effect. Values below the lower limit of quantification were set to the quantification limit for summary.
Time Frame: Day 4
Population: as for outcome 3
Measure: Geometric Mean (Standard Deviation); unit: Nanomoles per liter (nmol/L)
Arm/Group | Albiglutide 50 mg | Placebo
Number analyzed (Participants) | 20 | 21
Nanomoles per liter (nmol/L)
  0 hr, n=20, 21 | 1.095 (1.4141) | 0.836 (1.2694)
  1 hr, n=20, 21 | 1.616 (1.9504) | 0.993 (1.8530)
  1 hr 15 min, n=20, 21 | 1.630 (1.9941) | 1.053 (1.8949)
  1 hr 45 min, n=20, 21 | 0.786 (2.2046) | 0.517 (1.8094)
  2 hr, n=20, 20 | 0.723 (2.1648) | 0.484 (1.8073)
  2 hr 45 min, n=20, 21 | 0.362 (2.2903) | 0.275 (1.8736)
  3 hr, n=20, 21 | 0.309 (2.2762) | 0.255 (1.8769)
  3 hr 30 min, n=20, 21 | 0.152 (1.7438) | 0.138 (1.3718)
  3 hr 45 min, n=20, 21 | 0.140 (1.5595) | 0.128 (1.3047)
  4 hr 15 min, n=20, 21 | 0.105 (1.1483) | 0.101 (1.0589)
  4 hr 30 min, n=20, 21 | 0.100 (1.0000) | 0.100 (1.0000)
  4 hr 45 min, n=20, 21 | 0.100 (1.0000) | 0.100 (1.0000)
  5 hr, n=20, 21 | 0.105 (1.1483) | 0.103 (1.0821)
  5 hr 15 min, n=20, 21 | 0.118 (1.4512) | 0.120 (1.3662)
  5 hr 30 min, n=20, 21 | 0.141 (1.6701) | 0.138 (1.4534)

9. Secondary Outcome: Recovery Time of Plasma Glucose Levels to >=3.9 mmol/L (>=70 mg/dL) From the Hypoglycemic Clamp Level of 2.8 Nmol/L (50.4 mg/dL)
Description: The effect of albiglutide and placebo on the recovery time of plasma glucose levels to >=3.9 mmol/L (7>=0 mg/dL) from the hypoglycemic clamp level of 2.8 nmol/L (50.4 mg/dL) was calculated as the time in minutes between switching off of the insulin infusion and reaching the level of >=3.9 mmol/L (>=70 mg/dL). Censored values were censored at 70 minutes. The median and 95% confidence interval data are obtained from Kaplan-Meier estimates.
Time Frame: Day 4
Population: Pharmacodynamic Population
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Albiglutide 50 mg | Placebo
Number analyzed (Participants) | 20 | 21
Minutes | 35.00 [30.00 to 45.00] | 30.00 [25.00 to 40.00]

10. Secondary Outcome: Average Albiglutide Concentration on the Day of the Clamp Procedure
Description: Plasma samples were taken from participants at two time points on Day 4 (at 0 hours and 4 hours and 45 minutes post-dose) of Week 1 of the study for albiglutide study drug level analyses. The average concentration for each participant was calculated as the mean of the concentrations at 0 hours and 4 hours 45 minutes. The clamp procedure is a glucose-controlled insulin infusion system. Variable infusions of glucose are administered to achieve various glucose target levels. It is a way of quantifying insulin secretion and resistance.
Time Frame: Day 4
Population: Albiglutide Pharmacokinetic Population: all participants who had at least one sample to compute albiglutide exposure
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Albiglutide 50 mg | Placebo
Number analyzed (Participants) | 19 | 0
Nanograms per milliliter (ng/mL)
  Week 1, Day 4, 0 hours | 2110.5 (905.81) |
  Week 1, Day 4, 4 hours 45 minutes | 1968.7 (754.37) |
  Average Concentration | 2039.63 (826.584) |

11. Secondary Outcome: Number of Participants With Any Treatment-emergent Serious Adverse Event (SAE) and Treatment-emergent Non-serious Adverse Event (AE) During the Clamp Period
Description: Treatment-emergent AEs are defined as those with an onset on or after study drug administration. An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect.
Time Frame: From the time the participant consented to participate in the study through the end of the study, or the final follow-up visit for participants who discontinued active participation in the study (up to 8 study weeks)
Population: Safety Population: all participants who received one dose of albiglutide or placebo. The Safety Population was analyzed according to treatment received.
Measure: Number; unit: Participants
Arm/Group | Albiglutide 50 mg | Placebo
Number analyzed (Participants) | 22 | 22
Participants
  Any treatment-emergent non-serious AE | 9 | 10
  Any treatment-emergent SAE | 0 | 0

ADVERSE EVENTS:
Time Frame: SAEs and non-serious AEs were collected from the time the participant consented to participate in the study through the end of the study, or the final follow-up visit for participants who discontinued active participation in the study (up to 8 weeks).
Description: On-therapy SAEs and non-serious AEs (onset on or after the first day of study medication) were collected in members of the Safety Population, comprised of all randomly assigned study participants who received at least one dose of study medication.
Arm/Group | Albiglutide 50 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 3/22 | 4/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Albiglutide 50 mg (N=22) | Placebo (N=22)
Headache (Nervous system disorders) | 1 | 2
Gastroenteritis (Infections and infestations) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.